CLINICAL TRIAL: NCT04947293
Title: Effects of Yoga in the Rehabilitation of Stroke Patients With Chronic Sequelea: A Randomized Controlled Trial.
Brief Title: Yoga Among Stroke Patients With Chronic Sequelae
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital La Musse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-A03408-31
Record Dates: First submitted 2021-06-11; First posted 2021-07-01 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Chronic Stroke
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga Exercise (Experimental): Subjects in the experimental group will be invited to participate in 60-minute yoga sessions twice a week for 12 weeks. Each session will include postural (asanas), breathing (pranayama), and meditative exercises. They will be adapted to the physical possibilities of the patients with the help of accessories such as chairs, straps, blankets, blocks. One additional session (60 minutes) per week, in autonomy, at home, will be recommended and accompanied by a video support.
  Interventions: Other: Physical activity
- Fitness and mobility exercise (Active Comparator): Subjects in the control group will be invited to participate in more conventional exercise sessions, based on a fitness and mobility exercise (FAME) program, 60-minute per sessions twice a week for 12 weeks. One additional session (60 minutes) per week, in autonomy, at home, will be recommended and accompanied by a video support. The effectiveness of this program has already been demonstrated in previous studies.
  Interventions: Other: Physical activity

INTERVENTIONS:
Other: Physical activity — Both groups will practice a physical activity adapted to their motor skills. They will have two group sessions (maximum 5 people per group) in a face-to-face setting, and one independent session at home supported by a video, each week. These programs last 12 weeks, and will be supervised by the same person, a physiotherapist.

SUMMARY:
Stroke is a major health problem and can cause long-term disability. Among these sequelae, there are balance and mobility disorders, but also a higher rate of anxiety or depression disorders. This impairments impact activity of daily living, and social reintegration. That why the investigators need to explore options for long-term sustainable interventions that which takes into account the patient as a whole. In particular, regular physical activity is recommended, but it must be adaptable to the patient's impairments. Teaching yoga may be an interesting option. Indeed, yoga is a mind-body practice which become increasingly widespread in the world. Recent studies highlight positive effect of yoga for this population. However, the levels of evidence are limited, and new studies are needed.

Primary objective of the study is to demonstrate the non-inferiority of a therapeutic yoga program, compared to a conventional physical activity program, to improve balance of patients with chronic stroke sequelae.

Secondary objectives are to demonstrate the non-inferiority of the therapeutic yoga program in improving muscle strength and functional mobility, as well as its superiority in improving anxiety, depression, social reintegration and adherence to treatment.

DETAILED DESCRIPTION:
The investigators will conduct a single-blind randomised controlled trial to study the effectiveness of a yoga programme compared to a conventional adapted physical activity programme in improving balance in chronic post-stroke subjects. The primary hypothesis is that yoga is non-inferior to conventional physical activity in improving balance in chronic post-stroke patients. The secondary hypothesis is that yoga is non-inferior to conventional physical activity in improving muscle strength and functional mobility, but superior in improving anxiety, depression, social reintegration and treatment adherence.

The experiment will take place in Normandy (France), at several sites in order to maximise recruitment and minimise travel for participants. The statistical power study indicates that 42 patients per group would be required. Subjects will be randomly assigned to one of the following programmes: the YOG'AVC programme or the FAME programme. The first will involve yoga sessions with postural, respiratory, and meditative work. The second will involve more conventional exercise sessions, based on a Fitness and Mobility Exercise Program (FAME) designed for stroke survivors. Both programmes included two 60-minute group sessions per week, for 12 weeks, plus one weekly home-based session (with video or paper support). Patients will be assessed at three points in the study: before the experiment (T0), after the 12-week experiment (T1), and 3 months later (T2). The assessments will be carried out blind, using a protocol built around the International Classification of Functioning and Disability (ICF). The main criterion is balance, assessed by the Berg balance scale (0-56 point scale). The secondary outcomes will be assessed by: Timed Up and Go Test (timed task in seconds), 6-minute walk test (distance covered in meters), maximum isometric knee extension force with a manual dynamometer (newton), the activities-specific Balance Confidence Scale - Simplified (questionnaire in %), State-Trait Anxiety Inventory (2 questionnaires out of 80), Beck Depression Inventory (score out of 63), Reintegration to Normal Living Index (score out of 100). Adherence to the programme will be assessed by a logbook, between T0 and T1 by the number of group and individual sessions completed, and between T1 and T2 by the number of self-reported sessions.

ELIGIBILITY:
Inclusion Criteria:

* a minimum of six month elapsed time since stroke incidence
* present balance disorders (score between 21 and 51 on the Berg Balance Scale)
* ability to stand and walk at least 10 metres (with or without an assistance device)
* be affiliated to a social security system

Exclusion Criteria:

* under 18 years of age
* cognitive impairment assessed by a score of less than 4 on the 6-items Mini-Mental State Examination
* inability to understand the French language (to the point of not being able to answer questionnaires, or understand instruction)
* medical contraindication to the practice of a sport activity
* current and regular participation in a physical activity program
* Being deprived of liberty by a judicial or administrative decision,
* Receive psychiatric care,
* Be subject to a legal protection measure (guardianship, curatorship and safeguarding of justice),
* Being a pregnant, parturient or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-08-21 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Functional Balance | Baseline
  Berg Balance Scale : This test is used to quantitatively assess balance in older adults. In this 14-item scale, patients are asked to maintain positions and perform movement tasks of varying degrees of difficulty. Patients receive a score between 0 and 4 on their ability to respond to dimensions of balance. An overall score can be calculated from a total of 56. The higher the score, the better the balance. This scale has been found to be reliable, valid, and is the most commonly used clinical and research scale for assessing balance in stroke patients.
Functional Balance | Immediately after the intervention
  Berg Balance Scale : This test is used to quantitatively assess balance in older adults. In this 14-item scale, patients are asked to maintain positions and perform movement tasks of varying degrees of difficulty. Patients receive a score between 0 and 4 on their ability to respond to dimensions of balance. An overall score can be calculated from a total of 56. The higher the score, the better the balance. This scale has been found to be reliable, valid, and is the most commonly used clinical and research scale for assessing balance in stroke patients.
Functional Balance | 3 months follow-up
  Berg Balance Scale : This test is used to quantitatively assess balance in older adults. In this 14-item scale, patients are asked to maintain positions and perform movement tasks of varying degrees of difficulty. Patients receive a score between 0 and 4 on their ability to respond to dimensions of balance. An overall score can be calculated from a total of 56. The higher the score, the better the balance. This scale has been found to be reliable, valid, and is the most commonly used clinical and research scale for assessing balance in stroke patients.

SECONDARY OUTCOMES:
Functional mobility | Baseline
  Timed Up and Go Test : It is a test based on the performance of a functional task, where the subject must get up from a chair, walk 3 meters, turn around and return to a seat. The subject is timed during the execution and a score in seconds is established. The reliability and validity of this test was established in a chronic stroke population.
Functional mobility | Immediately after the intervention
  Timed Up and Go Test : It is a test based on the performance of a functional task, where the subject must get up from a chair, walk 3 meters, turn around and return to a seat. The subject is timed during the execution and a score in seconds is established. The reliability and validity of this test was established in a chronic stroke population.
Functional mobility | 3 months follow-up
  Timed Up and Go Test : It is a test based on the performance of a functional task, where the subject must get up from a chair, walk 3 meters, turn around and return to a seat. The subject is timed during the execution and a score in seconds is established. The reliability and validity of this test was established in a chronic stroke population.
Gait performance | Baseline
  The 6-minute walk test (TDM6) : an endurance test where the subject must walk for 6 minutes over the longest possible distance (score in meters). This test is reliable and valid for a chronic stroke population.
Gait performance | Immediately after the intervention
  The 6-minute walk test (TDM6) : an endurance test where the subject must walk for 6 minutes over the longest possible distance (score in meters). This test is reliable and valid for a chronic stroke population.
Gait performance | 3 months follow-up
  The 6-minute walk test (TDM6) : an endurance test where the subject must walk for 6 minutes over the longest possible distance (score in meters). This test is reliable and valid for a chronic stroke population.
Maximum isometric muscle strength of the knee extensors | Baseline
  Manual dynamometer (Microfet2®). Subject is seated, knees and hips bent at 90°. The dynamometer is placed on the anterior surface of the tibia, 5 cm from the malleoli, with a tip adapted to the surface being tested. The subject is invited to push against the resistance, as if stretching the leg, with all the force he or she can muster. The measurement is repeated 3 times, and the score (in Newton) is established by averaging the 3 trials. Hand-held dynamometry is a reliable and valid method for assessing muscle strength in a stroke population.
Maximum isometric muscle strength of the knee extensors | Immediately after the intervention
  Manual dynamometer (Microfet2®). Subject is seated, knees and hips bent at 90°. The dynamometer is placed on the anterior surface of the tibia, 5 cm from the malleoli, with a tip adapted to the surface being tested. The subject is invited to push against the resistance, as if stretching the leg, with all the force he or she can muster. The measurement is repeated 3 times, and the score (in Newton) is established by averaging the 3 trials. Hand-held dynamometry is a reliable and valid method for assessing muscle strength in a stroke population.
Maximum isometric muscle strength of the knee extensors | 3 months follow-up
  Manual dynamometer (Microfet2®). Subject is seated, knees and hips bent at 90°. The dynamometer is placed on the anterior surface of the tibia, 5 cm from the malleoli, with a tip adapted to the surface being tested. The subject is invited to push against the resistance, as if stretching the leg, with all the force he or she can muster. The measurement is repeated 3 times, and the score (in Newton) is established by averaging the 3 trials. Hand-held dynamometry is a reliable and valid method for assessing muscle strength in a stroke population.
Activities-specific Balance Confidence Scale - Simplified | Baseline
  This questionnaire consists of 16 questions that require the patient to assess his or her confidence that he or she will not lose balance while performing the cited activities. For each of the 16 activities, the patient is asked to rate their confidence from 0 (not at all confident) to 3 (very confident). The total score is given as a percentage. The reliability and validity of the French version of this questionnaire has been established.
Activities-specific Balance Confidence Scale - Simplified | Immediately after the intervention
  This questionnaire consists of 16 questions that require the patient to assess his or her confidence that he or she will not lose balance while performing the cited activities. For each of the 16 activities, the patient is asked to rate their confidence from 0 (not at all confident) to 3 (very confident). The total score is given as a percentage. The reliability and validity of the French version of this questionnaire has been established.
Activities-specific Balance Confidence Scale - Simplified | 3 months follow-up
  This questionnaire consists of 16 questions that require the patient to assess his or her confidence that he or she will not lose balance while performing the cited activities. For each of the 16 activities, the patient is asked to rate their confidence from 0 (not at all confident) to 3 (very confident). The total score is given as a percentage. The reliability and validity of the French version of this questionnaire has been established.
State Trait Anxiety Inventory | Baseline
  The 2 forms of the State Trait Anxiety Inventory (STAI, Form Y) will use to measure state anxiety (STAI-Y1) and trait anxiety (STAI-Y2).
  The 2 forms consist of 20 items each, which are rated on a 4-point Likert-type scale depending on how the participant feels at the moment in time for STAI-Y1 or how the participant feels generally for STAI-Y2. Higher scores are associated with increased symptoms of state or trait anxiety.
State Trait Anxiety Inventory | Immediately after the intervention
  The 2 forms of the State Trait Anxiety Inventory (STAI, Form Y) will use to measure state anxiety (STAI-Y1) and trait anxiety (STAI-Y2).
  The 2 forms consist of 20 items each, which are rated on a 4-point Likert-type scale depending on how the participant feels at the moment in time for STAI-Y1 or how the participant feels generally for STAI-Y2. Higher scores are associated with increased symptoms of state or trait anxiety.
State Trait Anxiety Inventory | 3 months follow-up
  The 2 forms of the State Trait Anxiety Inventory (STAI, Form Y) will use to measure state anxiety (STAI-Y1) and trait anxiety (STAI-Y2).
  The 2 forms consist of 20 items each, which are rated on a 4-point Likert-type scale depending on how the participant feels at the moment in time for STAI-Y1 or how the participant feels generally for STAI-Y2. Higher scores are associated with increased symptoms of state or trait anxiety.
Beck Depression Inventory | Baseline
  This self-questionnaire includes 21 items identifying symptoms and attitudes associated with depression. Each item is assessed on a severity scale ranging from 0 to 3, with a total score ranging from 0 to 63.The higher the score, the more severe the depression. The reliability and validity of the French version of this questionnaire has been established.
Beck Depression Inventory | Immediately after the intervention
  This self-questionnaire includes 21 items identifying symptoms and attitudes associated with depression. Each item is assessed on a severity scale ranging from 0 to 3, with a total score ranging from 0 to 63.The higher the score, the more severe the depression. The reliability and validity of the French version of this questionnaire has been established.
Beck Depression Inventory | 3 months follow-up
  This self-questionnaire includes 21 items identifying symptoms and attitudes associated with depression. Each item is assessed on a severity scale ranging from 0 to 3, with a total score ranging from 0 to 63.The higher the score, the more severe the depression. The reliability and validity of the French version of this questionnaire has been established.
Reintegration to Normal Living Index | Baseline
  This self-questionnaire was developed to quantitatively assess the degree to which individuals who have experienced a traumatic or disabling illness are able to reintegrate into normal social activities (e.g., recreational activities, movement in the community, and interactions with family and other relationships). It is composed of 11 declarative statements (e.g. I move around my home as much as I want), and the patient gives a score between 0 and 2 (yes, partially, no). The total score is between 0 and 22 points, a high score indicates low reintegration.
Reintegration to Normal Living Index | Immediately after the intervention
  This self-questionnaire was developed to quantitatively assess the degree to which individuals who have experienced a traumatic or disabling illness are able to reintegrate into normal social activities (e.g., recreational activities, movement in the community, and interactions with family and other relationships). It is composed of 11 declarative statements (e.g. I move around my home as much as I want), and the patient gives a score between 0 and 2 (yes, partially, no). The total score is between 0 and 22 points, a high score indicates low reintegration.
Reintegration to Normal Living Index | 3 months follow-up
  This self-questionnaire was developed to quantitatively assess the degree to which individuals who have experienced a traumatic or disabling illness are able to reintegrate into normal social activities (e.g., recreational activities, movement in the community, and interactions with family and other relationships). It is composed of 11 declarative statements (e.g. I move around my home as much as I want), and the patient gives a score between 0 and 2 (yes, partially, no). The total score is between 0 and 22 points, a high score indicates low reintegration.
Compliance during the program | During the intervention
  A percentage will be established according to the number of sessions actually performed compared to the number of planned sessions.
Compliance after the program | 3 months follow-up
  A percentage will be established based on the number of sessions actually completed compared to the number of sessions recommended.

CONTACTS AND LOCATIONS:
Overall Officials: Maxime Gilliaux, PhD, Principal Investigator — Hôpital La Musse
Locations (3):
- France (3):
  - City hall of Broglie, Broglie, Eure
  - City Hall of Corneville sur Risle, Corneville-sur-Risle
  - Hopital La Musse, Saint-Sébastien-de-Morsent

IPD SHARING:
Plan to Share IPD: No
The data collected will be anonymized, computerized and stored by Maxime GILLIAUX. Only the investigators will have access to the anonymized data in order to carry out the statistical work of this research.

REFERENCES:
- [Background] Green E, Huynh A, Broussard L, Zunker B, Matthews J, Hilton CL, Aranha K. Systematic Review of Yoga and Balance: Effect on Adults With Neuromuscular Impairment. Am J Occup Ther. 2019 Jan/Feb;73(1):7301205150p1-7301205150p11. doi: 10.5014/ajot.2019.028944. PMID 30839270
- [Background] Thayabaranathan T, Andrew NE, Immink MA, Hillier S, Stevens P, Stolwyk R, Kilkenny M, Cadilhac DA. Determining the potential benefits of yoga in chronic stroke care: a systematic review and meta-analysis. Top Stroke Rehabil. 2017 May;24(4):279-287. doi: 10.1080/10749357.2016.1277481. Epub 2017 Jan 19. PMID 28100160
- [Background] Edwards MK, Loprinzi PD. Comparative effects of meditation and exercise on physical and psychosocial health outcomes: a review of randomized controlled trials. Postgrad Med. 2018 Mar;130(2):222-228. doi: 10.1080/00325481.2018.1409049. Epub 2017 Nov 27. PMID 29164993